CLINICAL TRIAL: NCT02665754
Title: The Efficacy and Adverse Effect of Intralymphatic Immunotherapy With Tyrosine S®, Allergen Extract for Immunotherapy, in Patients With Allergic Rhinitis Induced by House Dust Mite, Dog, and Cat Allergen
Brief Title: Intralymphatic Immunotherapy for House Dust Mite, Dog, and Cat Allergy Using Tyrosine S® in Allergic Rhinitis
Acronym: ILIT-T
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Korea Research Foundation (Other)
Responsible Party: Principal Investigator, Sangmin Lee, MD, Assistant Professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBIRB2016-002
Record Dates: First submitted 2016-01-10; First posted 2016-01-28 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Injection, intralymphatic; Immunotherapy; Dermatophagoides farinae; Dermatophagoides pteronyssinus; Dogs; Cats
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Saline Solution; Interleukin-13

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active group (Experimental): In active group, extract of causal allergen will be injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval.
  Interventions: Biological: ILIT with extract of causal allergen; Drug: Rescue medication for allergic rhinitis
- Placebo group (Placebo Comparator): In placebo group, normal saline will be injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval.
  Interventions: Biological: ILIT with normal saline; Drug: Rescue medication for allergic rhinitis

INTERVENTIONS:
Biological: ILIT with extract of causal allergen — 0.5 ml of allergen extract from D. farinae, D. pteronyssinus, cat, and/or dog for allergen specific immunotherapy (Tyrosine S, Allergy Therapeutic, UK) will be injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval.
  Other Names: Active ILIT
  Arms: Active group
Biological: ILIT with normal saline — 0.5 ml of normal saline will be injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval.
  Other Names: Placebo ILIT
  Arms: Placebo group
Drug: Rescue medication for allergic rhinitis — Subjects are requested to administer oral antihistamine (cetirizine) or nasal glucocorticosteroid (ciclesonide) as rescue medication for allergic rhinitis in accordance with severity and frequency of allergic rhinitis symptoms according to Allergic Rhinitis and its Impact on Asthma (ARIA) guideline.
  Other Names: Rescue medication

SUMMARY:
The investigators will perform double-blinded placebo-controlled randomized clinical trial which evaluates the efficacy and safety of allergen-specific intralymphatic immunotherapy (ILIT) for allergens including Dermatophagoides farinae (Df), Dermatophagoides pteronyssinus (Dp), cat, and dog that are sensitized and provoke rhinitis-related symptoms in patients with allergic rhinitis (AR), using allergen extracts for allergen-specific immunotherapy (Tyrosine S, Allergy Therapeutic, West Sussex, UK).

DETAILED DESCRIPTION:
After informed consent, subjects will be randomly assigned to ILIT group or placebo group in double-blind manner. In both group, causal allergen or placebo will be injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval. In ILIT group, initial dose of allergen will be 1,000-fold diluted solution from maximal concentration of allergen extract for subcutaneous immunotherapy (Tyrosine S, Allergy Therapeutic, West Sussex, UK) in volume of 0.1ml. If skin is highly reactive in skin prick test, the initial dose will be 10-fold dilution from maximal concentration where diameter of wheal is less than that of histamine. After the first dose, allergen concentration will be escalated 3-fold at second dose, and 10-fold at third dose if there are no (or mild) local or systemic hypersensitivity reaction. The allergen concentration will not change at second or third dose if there is moderate local or systemic reaction. The allergen concentration will decrease by 10 or 100-fold from previous concentration or further injection will be held if there is severe local or systemic reaction after sufficient explanation and discussion with subjects.

The investigators will evaluate allergic rhinitis symptom score before and 4, 12 months after the initial treatment. Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) and Sino-Nasal Outcome Test (SNOT-20) will be used. Visual analogue scale (VAS) of symptoms including rhinorrhea, sneezing, nasal obstruction, postnasal drip, eye/nose/ear/palate itching, dyspnea, wheezing, chest discomfort as well as urticaria, angioedema, and itching on exposed skin during exposure to causal allergen in daily life will be also evaluated. Skin prick test (SPT), intradermal test (IDT), blood sampling for serum total immunoglobulin E (IgE), allergen-specific IgE, and allergen-specific immunoglobulin G4 (IgG4), nasal lavage for Th1, Th2, and Treg cytokines, and nasal provocation test (NPT) with Df and/or Dp allergen (in subjects whose AR symptoms are provoked by Df and/or Dp) will be also performed before and 4, 12 months after the initial treatment. In addition, the investigators evaluated the change of subjects' recognition of causal allergens, their avoidance, and AIT during this study. Using VAS, subjects were requested to score the rate of agreement with "Allergen provokes allergic symptoms in daily life", "Allergen avoidance can reduce allergic symptoms", "Allergen-specific Immunotherapy (AIT) can reduce allergic symptoms", "I can pay 50,000 Korean Won (KRW)/month for allergen avoidance", "I can pay 100,000 KRW/month for allergen avoidance", "I can pay 200,000 KRW/month for allergen avoidance", "I can pay 150,000 KRW for each injection of ILIT", "I can pay 300,000 KRW for each injection of ILIT", "I can pay 600,000 KRW for each injection of ILIT" before and after SPT/IDT, after NPT, 4 months and 1 year after ILIT.

Adverse events will be recorded and graded according to Muller classification and Ring and Meissner classification.

ELIGIBILITY:
Inclusion Criteria:

We enrolled subjects who suffered from AR, symptoms of which were provoked by Dp, Df, dog, and/or cat allergen. Concretely, two inclusion criteria should be met.

1. Sensitization should be verified by skin prick test and the level of serum specific IgE measured by ImmunoCAP® (Thermo Fisher Scientific, Uppsala, Sweden).
2. Subjects should complain of AR symptoms during exposure of house dust, dog and/or cat in daily life.

Exclusion Criteria:

1. Uncontrolled or severe asthma according to Global Initiative of Asthma (GINA) guideline including a case in which forced expiratory volume in 1 s (FEV1) was less than 50% of predicted value
2. Significant cardiovascular, hepatic, renal, hematologic, oncologic, or infectious diseases
3. Administration of beta blocker, angiotensin converting enzyme inhibitor, tricyclic antidepressant, immunosuppressant including systemic glucocorticosteroid within last 2 weeks
4. AR caused by other perennial or seasonal allergen
5. Prior history of allergen-specific immunotherapy
6. Rejection or low compliance,
7. Pregnancy or lactation
8. Vulnerable volunteer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
RQLQ | 4 months after the day of first injection of ILIT
  Rhinoconjunctivitis Quality of Life Questionnaires

SECONDARY OUTCOMES:
SNOT-20 | before and 4, 12 months after the day of first injection of ILIT
  Sinonasal Outcome Test-20
Allergic symptoms provoked by causal allergen in daily life | before and 4, 12 months after the day of first injection of ILIT
  Rates scored by subjects using visual analogue scale regarding allergic symptoms provoked by causal allergen in daily life
Rhinitis symptom in nasal provocation test | before and 4, 12 months after the day of first injection of ILIT
  Rhinitis symptom (visual analogue scale: 0~100) during nasal provocation test with allergen of D. farinae and/or D. pteronyssinus in subjects in whom D. farinae and/or D. pteronyssinus is causal allergen.
Skin reactivity in skin prick test | before and 4, 12 months after the day of first injection of ILIT
  Mean diameters of wheal caused by 1- to 10^7- fold dilution of causal allergen in skin prick test and their allergen histamine ratio
Skin reactivity in intradermal test | before and 4, 12 months after the day of first injection of ILIT
  Mean diameters of wheal caused by 10^2- to 10^7- fold dilution of causal allergen in intradermal test and their allergen saline ratio
Serum total IgE level | before and 4, 12 months after the day of first injection of ILIT
  Serum total IgE level using ImmunoCAP (Thermo Fisher Scientific, Uppsala, Sweden)
Allergen-specific IgE for causal allergen | before and 4, 12 months after the day of first injection of ILIT
  Allergen-specific IgE for causal allergen of D. farinae, D. pteronyssinus, cat, and/dog using ImmunoCAP (Thermo Fisher Scientific, Uppsala, Sweden)
Cytokines in nasal lavage fluid before and after nasal provocation test | before and 4, 12 months after the day of first injection of ILIT
  Cytokines of Th1, Th2, and Treg immunity including interleukin-4 (IL-4), IL-5, IL-10, IL-12, IL-13, interferon-gamma (IFN-g), and tumor growth factor-beta (TGF-b) in nasal lavage fluid
Subjects' score (0~100) regarding agreement to "Allergen provokes allergic symptoms in daily life" | before skin prick test / intradermal test, nasal provocation test, and 4, 12 months after the day of first injection of ILIT
  Subjects' score regarding agreement to "Allergen provokes allergic symptoms in daily life" using visual analogue scale (0~100).
Subjects' score (0~100) regarding agreement to "Allergen avoidance can reduce allergic symptoms" | before skin prick test / intradermal test, nasal provocation test, and 4, 12 months after the day of first injection of ILIT
  Subjects' score regarding agreement to "Allergen avoidance can reduce allergic symptoms" using visual analogue scale (0~100).
Subjects' score (0~100) regarding agreement to "Allergen-specific immunotherapy can reduce allergic symptoms" | before skin prick test / intradermal test, nasal provocation test, and 4, 12 months after the day of first injection of ILIT
  Subjects' score regarding agreement to "Allergen-specific immunotherapy can reduce allergic symptoms" using visual analogue scale (0~100).
Willingness to pay for allergen avoidance | before skin prick test / intradermal test, nasal provocation test, and 4, 12 months after the day of first injection of ILIT
  Agreement% scored by subjects using visual analogue scale to "I am willing to pay 50,000, 100,000 or 200,000 Korean Won per month for allergen avoidance"
Willingness to pay for intralymphatic immunotherapy | before skin prick test / intradermal test, nasal provocation test, and 4, 12 months after the day of first injection of ILIT
  Agreement% scored by subjects using visual analogue scale to "I am willing to pay 150,000, 300,000 or 600,000 Korean Won for each injection of intralymphatic immunotherapy"
Nasal mucosal inflammation | before and 4, 12 months after the day of first injection of ILIT
  Inflammatory cell count in nasal mucosal biopsy (/high power field, x400)
RQLQ | 12 months after the day of first injection of ILIT
  Rhinoconjunctivitis Quality of Life Questionnaires
Nasal cavitary volume decrease in nasal provocation test | before and 4, 12 months after the day of first injection of ILIT
  Nasal cavitary volume decrease (basal%) measured by acoustic rhinometry during nasal provocation test with allergen of D. farinae and/or D. pteronyssinus in subjects in whom D. farinae and/or D. pteronyssinus is causal allergen.
Allergen-specific IgG4 for causal allergen | before and 4, 12 months after the day of first injection of ILIT
  Allergen-specific IgG4 for causal allergen of D. farinae, D. pteronyssinus, cat, and/dog using ImmunoCAP (Thermo Fisher Scientific, Uppsala, Sweden)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy. Curr Opin Allergy Clin Immunol. 2009 Dec;9(6):537-43. doi: 10.1097/ACI.0b013e3283310ff7. PMID 19680119
- [Background] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy: from the rationale to human applications. Curr Top Microbiol Immunol. 2011;352:71-84. doi: 10.1007/82_2011_133. PMID 21725898
- [Background] Kundig TM, Johansen P, Bachmann MF, Cardell LO, Senti G. Intralymphatic immunotherapy: time interval between injections is essential. J Allergy Clin Immunol. 2014 Mar;133(3):930-1. doi: 10.1016/j.jaci.2013.11.036. Epub 2014 Jan 15. No abstract available. PMID 24439076
- [Background] Johansen P, Kundig TM. Intralymphatic immunotherapy and vaccination in mice. J Vis Exp. 2014 Feb 2;(84):e51031. doi: 10.3791/51031. PMID 24513675
- [Background] Graf N, Dinkel B, Rose H, Hothorn LA, Gerhard D, Johansen P, Kundig TM, Klimek L, Senti G. A critical appraisal of analyzing nasal provocation test results in allergen immunotherapy trials. Rhinology. 2014 Jun;52(2):137-41. doi: 10.4193/Rhino13.145. PMID 24932625
- [Background] Zaleska A, Eiwegger T, Soyer O, van de Veen W, Rhyner C, Soyka MB, Bekpen C, Demiroz D, Treis A, Sollner S, Palomares O, Kwok WW, Rose H, Senti G, Kundig TM, Ozoren N, Jutel M, Akdis CA, Crameri R, Akdis M. Immune regulation by intralymphatic immunotherapy with modular allergen translocation MAT vaccine. Allergy. 2014 Sep;69(9):1162-70. doi: 10.1111/all.12461. Epub 2014 Jul 12. PMID 24934402
- [Background] Senti G, Kundig TM. Intralymphatic immunotherapy. World Allergy Organ J. 2015 Mar 7;8(1):9. doi: 10.1186/s40413-014-0047-7. eCollection 2015. PMID 25780493
- [Background] Hjalmsdottir A, Wackerle-Men Y, Duda A, Kundig TM, Johansen P. Dosing intervals in intralymphatic immunotherapy. Clin Exp Allergy. 2016 Mar;46(3):504-7. doi: 10.1111/cea.12657. No abstract available. PMID 26470052
- [Result] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Result] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Result] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268
- [Result] Witten M, Malling HJ, Blom L, Poulsen BC, Poulsen LK. Is intralymphatic immunotherapy ready for clinical use in patients with grass pollen allergy? J Allergy Clin Immunol. 2013 Nov;132(5):1248-1252.e5. doi: 10.1016/j.jaci.2013.07.033. Epub 2013 Sep 13. No abstract available. PMID 24035151
- [Result] Patterson AM, Bonny AE, Shiels WE 2nd, Erwin EA. Three-injection intralymphatic immunotherapy in adolescents and young adults with grass pollen rhinoconjunctivitis. Ann Allergy Asthma Immunol. 2016 Feb;116(2):168-70. doi: 10.1016/j.anai.2015.11.010. Epub 2015 Dec 17. No abstract available. PMID 26706294
- [Derived] Park HJ, Kim SH, Shin YS, Park CH, Cho ES, Choi SJ, Park SH, Jung JH, Kang IG, Lee MS, Kim DW, Lee SM, Yang MS, Lee SP. Intralymphatic immunotherapy with tyrosine-adsorbed allergens: a double-blind, placebo-controlled trial. Respir Res. 2021 Jun 4;22(1):170. doi: 10.1186/s12931-021-01766-0. PMID 34088322